CLINICAL TRIAL: NCT04008459
Title: WiSPA: Walking and Balance Related to Sagittal Spinal Posture and Alignment
Brief Title: Walking and Balance Related to Sagittal Spinal Posture Alignment
Acronym: WiSPA
Status: Terminated | Type: Observational
Why Stopped: Recruitment no longer viable as spinal classes were stopped due to the COVID-19 situation.
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 14031
Record Dates: First submitted 2019-06-27; First posted 2019-07-05 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-07

CONDITIONS: Hyperkyphosis; Walking, Difficulty; Balance; Distorted; Spinal Disease; Osteoporosis; Spine Degeneration
MeSH Terms: conditions — Kyphosis; Mobility Limitation; Spinal Diseases; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Degenerative musculoskeletal spinal conditions: Participants are included who are enrolled in a 6-week physiotherapy exercise class aimed at improving function in people with degenerative spinal conditions.
  Interventions: Other: Therapeutic exercise class

INTERVENTIONS:
Other: Therapeutic exercise class — Physiotherapy exercise class includes education, stretching, strengthening, posture and balance interventions.

SUMMARY:
This study aims to improve understanding of the relationship between spinal alignment and walking and balance in people who have degenerative spinal conditions.

DETAILED DESCRIPTION:
This prospective cohort study will include people who are attending physiotherapy to address a degenerative spinal condition and measure them longitudinally. The investigators will measure spinal alignment, walking capacity and pattern, dynamic balance, and back muscle strength along with self-reported measures that reflect the person's functional self-efficacy, quality of life, and general health. Physical and self-reported outcome measures will be assessed at baseline before the physiotherapy-led exercise class commences, after completion at 6 weeks, and 6 months post baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participant is diagnosed with a degenerative spinal condition.
* Participant is willing and able to give informed consent for participation in the study.
* Men and women aged 18 years or older.
* Participant is able to understand and participate safely in a physiotherapy measurement assessment.
* Participant is enrolled in physiotherapy.

Exclusion Criteria:

* Participant is unable to stand independently.
* Participant has a neurological condition which alters motor function and/or postural control.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with a degenerative spinal condition who have been referred to outpatient physiotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-04-06 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Change in sagittal spinal alignment | 6 weeks post-baseline
  Alignment of the spine in the sagittal plane measured by a surface topography method

SECONDARY OUTCOMES:
Sagittal spinal alignment | 6 months
  Alignment of the spine in the sagittal plane measured by a surface topography method
2 minute walk test | 6 weeks and 6 months
  Distance walked in 2 minutes to measure exercise capacity
Gait analysis | 6 weeks and 6 months
  Spatiotemoral gait parameters measured using inertial measurement units
Tragus to wall distance | 6 weeks and 6 months
  Forward posture measurement using the distance from the ear to the wall
Four Square Step Test | 6 weeks and 6 months
  Dynamic balance test involving multidirectional stepping over obstacles
Timed loaded standing test | 6 weeks and 6 months
  Measurement of back extensor muscle strength and endurance
36-item Short Form Health Survey (SF-36) | 6 weeks and 6 months
  Health survey measuring aspects of quality of life. The questionnaire contains 36 questions which form 8 subscales: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health. Each question is directly transformed into a 0-100 scale with the lower the score the more disability.
Visual analogue pain scale | 6 weeks and 6 months
  Measurement of pain in a participant's back. The scale is along a horizontal 10 cm line with markings from 0 to 10, 0 indicating no pain and 10 indicating the worst pain imaginable.
Activities-specific Balance Confidence Scale | 6 weeks and 6 months
  Questionnaire measuring balance confidence in various situations. It contains 16 questions in which participants rate their confidence in performing the activities on a scale from 0-100, 0 representing no confidence and 100 representing complete confidence. The total score is calculated to be on a similar 0 to 100 scale.
Modified gait efficacy scale | 6 weeks and 6 months
  Questionnaire measuring walking confidence and self-efficacy. Each of the 10 items is scored on a 10-point Likert scale with 1 representing no confidence and 10 representing complete confidence. The total score ranges from 10-100.
Sagittal spinal alignment | Within 2 weeks of baseline
  Reliability re-test of alignment of the spine in the sagittal plane measured by a surface topography method

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hannink, DPT, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford, Oxon, United Kingdom